CLINICAL TRIAL: NCT02491424
Title: Direct Skeletal Fixation of Prosthetic Limbs Following Trans- Femoral Amputation - Study of an Intraosseous Transcutaneous Amputation Prosthesis (ITAP)
Brief Title: Intraosseous Transcutaneous Amputation Prosthesis
Acronym: (ITAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-01
Record Dates: First submitted 2015-06-15; First posted 2015-07-08 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2016-04

CONDITIONS: Traumatic Amputation of Lower Extremity
Keywords: Osseointegration; Direct skeletal attachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fixation of ITAP to lower limb amputees. (Experimental): Direct skeletal fixation of ITAP to lower limb amputees. 20 patients in the study will be fitted with Intraosseous Transcutaneous Amputation Prosthesis.
  The device has been designed to be surgically implanted in a one stage procedure.
  Interventions: Device: Direct skeletal fixation of ITAP to lower limb amputees.

INTERVENTIONS:
Device: Direct skeletal fixation of ITAP to lower limb amputees. — Intraosseous Transcutaneous Amputation Prosthesis (ITAPTM) fitting. The core ITAP™ design comprises of three discrete sections, the proximal section, which is the intramedullary stem secured into the medullary canal, the soft tissue integration flange and the transcutaneous component that passes through the skin.

SUMMARY:
Direct Skeletal Fixation of Prosthetic Limbs Following Trans-Femoral Amputation - Study of an Intraosseous Transcutaneous Amputation Prosthesis (ITAPTM).

DETAILED DESCRIPTION:
The core ITAP™ design comprises of three discrete sections, the proximal section, which is the intramedullary stem secured into the medullary canal, the soft tissue integration flange and the transcutaneous component that passes through the skin. The device has been designed to be surgically implanted in a one stage procedure. In greater detail:

Intra-medullary stem - this component is designed to match the natural shape of the canal and is designed using the same principles established and used for the fixation of massive endo-prosthetic replacements. In certain cases a hydroxyapatite ceramic (CaPO4) coating is used, providing enhanced uncemented fixation. In other cases, depending on the geometry of the intramedullary canal, the stem can be fixed in place using acrylic bone cement.

ELIGIBILITY:
Inclusion Criteria:

* Trans-femoral amputation
* 6 months or more attempted prosthetic rehabilitation (use of walking aids not relevant)
* Between the ages of 18 to 60 inclusive
* Length of stump: Sufficient bony stock for bony integration (at the investigator's discretion) and sufficient clearance (at the investigator's discretion) from medial joint line to accommodate failsafe device/ adaptor and knee mechanism
* Suitable soft tissues to perform the operative procedure
* Flexion Deformity (FFD) at hip no more than 15°
* Normal range of flexion and adduction other than FFD
* Oxford Grade 4 muscle power in all groups around hip
* Normal contralateral leg function
* Psychologically suitable (as deemed by screening process)
* Sufficient standard of English to understand the Patient Information Sheet and general study requirements
* Ability to understand and comply with study requirements - notably study timelines and additional clinic visits
* Patients willing to take part in the study and sign the Informed Consent form

Exclusion Criteria:

* Radiotherapy to target limb at any time
* Chemotherapy within the preceding 12 months
* Cognitive impairment likely to affect participation
* Pre-existing ipsilateral hip pathology
* Limited cardiorespiratory reserve / inability to walk at normal pace
* Any significant co-morbidity that, in the investigator's opinion, is likely to affect outcome (e.g. osteoporosis, heart disease, peripheral vascular disease, obesity or unrelated cancer)
* Any co-morbidity in the contra-lateral leg that precludes walking
* Any significant previous infection within the previous 12 months, such as apical stump sepsis or dental sepsis
* MRSA
* Using another silver-dosed medical device/treatment
* Patients with hypersensitivity to silver
* Concurrent medico-legal proceedings taking place
* Patients currently included in other clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Adhesion check in the skin surrounding the ITAP | 12 month post surgery
  Skin reaction assessment reviews the adhesion to the Implant at surface layer
Assessment of skin colour surrounding the ITAP | 12 month post surgery
  Skin reaction assessment reviews the skin colour
Measuring temperature of the skin surrounding the ITAP | 12 month post surgery
  Skin reaction assessment reviews the temperature of the skin surrounding the ITAP and compares it to the other leg
Condition of the skin surrounding the ITAP | 12 month post surgery
  Skin reaction assessment reviews the presence of exudate
Pain at the end of stump | 12 month post surgery
  Skin reaction assessment reviews the pain in the skin area surrounding the ITAP
Swelling of the skin around the ITAP | 12 month post surgery
  Skin reaction assessment reviews the swelling around the ITAP

SECONDARY OUTCOMES:
Radiographic assessment to measure osseointegration | 18 month post surgery
  Radiographic assessments to measure osseointegration
Radiographic assessments to measure fixation of the ITAP | 18 month post surgery
  Radiographic assessments to measure fixation of the ITAP
Microbiological assessment of the stump by standard microbiological screen. | 18 month post surgery
  Microbiological assessment of the stump by standard microbiological screen. Data will only be recorded in the CRF in the event of an infection.
Calculate QTFA to measure quality of life | 18 month post surgery
  General quality of life through Q-TFA ( Questionnaire for persons with a transfemoral amputation)
Calculate SIGAM to measure Limb specific mobility | 18 month post surgery
  Limb specific measure of mobility through the SIGAM mobility grades
Gait analysis at 18 months to measure mobility | 18 month post surgery
  Gait analysis in patients where appropriate and possible (this data will not be collected in the CRF)
Subjective Qualitative Interview at 18 months to assess patient outcome | 18 month post surgery
  A voluntary short one hour interview at the end of the study to discuss practical and emotional aspects of the process
Assessment of adverse events throughout the clinical trial | 18 month post surgery
  Device-related and procedure-related complications will be analysed to assess device safety.

CONTACTS AND LOCATIONS:
Overall Officials: Mr Robert Grimer, Principal Investigator — ROH
Locations (2):
- United Kingdom (2):
  - Royal Orthopaedic, Birmingham
  - Royal National Orthopaedic Hospital, Stanmore